CLINICAL TRIAL: NCT07232667
Title: Healthy Taiwan Cultivation Plan: Building an Active-ageing Lifestyle in Rural Taiwan Through Integrating Novel Healthcare Technology - From Mitigating Digital and Health Literacy Gap, Establishing a Mobile Interactive Pro-active-ageing Information Platform, to Exploring Multi-dimensional Digital Biomarkers of Ageing
Brief Title: Digital Technology for Active and Healthy Ageing in Taiwan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Principal Investigator, Ta-wei Guu, Consultant Psychiatrist, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH114-REC3-134
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Healthy Aging; Digital Health Literacy
Keywords: Elderly people; Wearable technology; Digital health literacy; Healthy aging; Health literacy; Digital gap; Digital biomarkers

STUDY DESIGN:
Intervention Model Description: single arm interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Promotion through Wearable and Mobile Technology (Experimental): Participants will join a community-based health program integrating wearables, mobile health platforms, and structured education to promote active lifestyles, enhance health literacy, and collect longitudinal data in older adults in rural Taiwan.
  Participants will:
  1. Wear a research-grade wrist actigraphy device (GeneActiv) to record activity, sleep, and light exposure for ≥2 weeks.
  2. Use the iMED mobile app (NHRI, Taiwan) for feedback, health education, and medication tracking.
  3. For participants with limited mobility, use an under-mattress iCue sensor to monitor respiration and movement.
  4. Attend Aging Well Taiwan sessions based on the WHO ICOPE framework.
  5. Provide baseline and follow-up blood samples for dementia-related biomarkers (Tau, Aβ, NfL) and APOE genotyping.
  Interventions: Device: Geneactiv; Behavioral: iMED Mobile Health Platform; Device: iCue; Behavioral: Aging Well Taiwan; Biological: Blood Biomarker Sampling

INTERVENTIONS:
Device: Geneactiv — Participants will wear a research-grade actigraphy device (Geneactiv original, developed by Activinsights UK) on the non-dominant wrist for at least two consecutive weeks to continuously record physical activity, sleep-wake patterns, and light exposure. The visualised results will be presented to the participants to motivate their behavioural change.
Behavioral: iMED Mobile Health Platform — Participants will use the "iMED" mobile application developed by the National Health Research Institutes in Taiwan (https://www.nhri.imed-health.com/). The platform provides personalized health education, medication reminders, AI-driven feedback on wearable data, and links to Taiwan's National Health Insurance health records.
Device: iCue — A non-invasive smart mat (iCue) placed under the mattress continuously monitors respiration rate, movement, and sleep parameters in participants with limited mobility.
Behavioral: Aging Well Taiwan — Participants will attend a community-based educational course adapted from Singapore's "Aging Well" framework, covering physical activity, diet, cognitive health, and digital literacy. The program follows the WHO Integrated Care for Older People (ICOPE) model and supports active aging and social participation.
Biological: Blood Biomarker Sampling — Participants will provide venous blood samples at baseline and follow-up visits for analysis of dementia-related biomarkers, including total Tau, phosphorylated Tau 181 (pT181), phosphorylated Tau 217 (pT217), amyloid beta 1-40 (Aβ40), amyloid beta 1-42 (Aβ42), and neurofilament light chain (NfL), as well as apolipoprotein E (APOE) genotyping.

SUMMARY:
Taiwan is entering a super-aged society in 2025, with more than 20% of the population aged 65 years or older. This rapid demographic shift, combined with increasing rates of chronic diseases, frailty, and dementia, has created growing challenges for healthcare and caregiving systems. Yunlin County, particularly its coastal region, has been one of Taiwan's earliest super-aged areas, showing higher rates of diabetes (10.5%), hypertension (28%), hyperlipidemia (26%), dementia (8%), and depression (12%) compared with national averages. Lifestyle factors such as tobacco (30%), betel nut (8%), and alcohol (15%) use are also more prevalent among local residents.

From 2022 to 2024, health screenings at CMU Beigang Hospital revealed a 36.1% abnormality rate among 12,222 visits, while another 5,965 assessments from the county's ICOPE program showed similarly high rates. Many older adults, particularly retired agricultural and fishing workers, experience sedentary lifestyles and polypharmacy-related risks, which worsen frailty, insomnia, depression, and cognitive decline. Low general and digital health literacy further limits their ability to adopt preventive behaviors, forming a vicious cycle between poor health and aging.

To address these challenges, the Ministry of Health and Welfare launched the "Healthy Taiwan Cultivation Plan." In alignment with this initiative, this project-led by CMU Beigang Hospital in collaboration with the National Health Research Institutes-aims to develop a wearable- and mobile-based health promotion model for rural older adults. The study will integrate research-grade actigraphy (Geneactiv), a mobile health platform ("iMED"), and the in-bed sensor iCue to monitor behavior, promote active aging, and enhance health and digital literacy. Ultimately, this project seeks to establish Taiwan's first integrated digital aging database and identify digital biomarkers for predicting cognitive and functional decline in older adults.

DETAILED DESCRIPTION:
This single-arm interventional study aims to develop a wearable and mobile health-based model to improve health and digital literacy among older adults living in rural Taiwan. The study focuses on Yunlin County, one of Taiwan's earliest super-aged regions, where chronic diseases, frailty, and dementia are highly prevalent. The project combines community-based interventions with continuous monitoring using wearable and digital tools to promote active aging and reduce health disparities.

The intervention integrates a research-grade wearable actigraphy device (Geneactiv), an AI-supported mobile health platform (iMED), and a smart in-bed sensor (iCue). These tools will continuously monitor physical activity, sleep patterns, and physiological parameters, while also providing real-time feedback and personalized health education. In addition, the "Aging Well Taiwan" program and the World Health Organization's Integrated Care for Older People (ICOPE) framework will be used to strengthen both health literacy and digital literacy among participants.

Phase I (2025-2026):

The first phase will establish baseline data and evaluate the feasibility, usability, and acceptability of wearable and mobile tools in community settings. Participants will wear GeneActiv devices for at least two weeks, complete ICOPE assessments, and provide blood samples for dementia-related biomarkers, including total Tau, phosphorylated Tau 181 (pT181), phosphorylated Tau 217 (pT217), amyloid beta 1-40 (Aβ40), amyloid beta 1-42 (Aβ42), and neurofilament light chain (NfL), as well as apolipoprotein E (APOE) genotyping. Validated questionnaires will be used to assess health literacy, digital literacy, and lifestyle factors.

Phase II (2027-2029):

The second phase will implement a single-arm intervention integrating the mobile health platform with wearable and sensor data. Participants will be followed up every three months to track changes in activity, sleep, medication use, mental well-being, and behavioral outcomes. Quantitative data will be analyzed using GGIR, R, and SPSS software, while qualitative interviews will explore usability, user satisfaction, and behavioral changes related to technology use.

This study will establish Taiwan's first integrated digital aging database that merges wearable, behavioral, and biological data. Through collaboration with international partners such as the RADAR-AD consortium, the project aims to identify digital phenotypes and biomarkers associated with cognitive and functional decline. Ultimately, the study aims to establish a sustainable, evidence-based, and technology-supported model that promotes healthy aging and improves well-being among older adults in rural communities.

ELIGIBILITY:
Inclusion Criteria:

1. Currently living or receiving care in a stable environment for at least four weeks prior to enrollment:

   * For community-based participants: must have resided at the same address for ≥4 weeks.
   * For day-care participants: must have attended activities at the same dementia or elderly day-care center for ≥4 weeks.
2. Able and willing to participate in the study procedures.
3. Informed consent must be obtained before participation.

   * If the participant's cognitive function has declined to a level that prevents self-consent, written consent will be obtained from a legally authorized representative or primary caregiver.

Exclusion Criteria:

1. Unstable physical or psychological condition that makes participation unsafe, as determined by a clinical investigator - e.g., acute delirium or current respiratory infection (including COVID-19).
2. Any known allergy or skin sensitivity to the materials used in the Geneactiv actigraphy device or iCue sensor pad.
3. Any other medical, neurological, or behavioral condition deemed unsuitable for participation by the study physician.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Activity-Sleep Pattern Regularity | Baseline to 36 months.
  Mean daily activity counts, sleep-wake cycles, and circadian rhythm stability will be assessed using Geneactiv and iCue in-bed sensors.
  Variables include total activity counts, sleep duration, sleep efficiency, wake after sleep onset (WASO), daytime napping, light exposure amount and timing, M5/L5 (five hours of highest/lowest activity), mean sleep midpoint (MSA), intra-daily variability (IV), inter-daily stability (IS), and Sleep Regularity Index (SRI).
  Data will be analyzed using the open-source GGIR algorithm and R software to evaluate individual day-night rhythm stability and longitudinal changes.
Integrated Care for Older People (ICOPE) Function Assessment | Baseline to 36 months.
  As assessed using the WHO Integrated Care for Older People (ICOPE) screening tool, covering six domains: cognition, mobility, nutrition, vision, hearing, and mood. Scores are classified as "declined" or "maintained" function for each domain. Higher functional integrity across domains indicates better overall health status.
Biomarkers for Cognitive and Functional Decline | Two time points - baseline (before intervention) and end of study (month 36).
  Venous blood samples (10 mL) will be collected to measure total Tau, phosphorylated Tau 181 (pT181), phosphorylated Tau 217 (pT217), amyloid beta 1-40 (Aβ40), amyloid beta 1-42 (Aβ42), and neurofilament light chain (NfL) using validated immunoassays.
  APOE genotyping will be performed once at baseline. These blood-based biomarkers will be correlated with digital device-derived metrics (SRI, IS, IV) and cognitive outcomes to explore their potential as predictors of cognitive decline.
Qualitative Evaluation of Feasibility and User Experience | Baseline to 36 months (post-intervention qualitative evaluation).
  Semi-structured interviews and focus groups will be conducted with participants and caregivers to explore usability, satisfaction, and perceived benefits of the Geneactiv wearable, iCue in-bed sensor, and iMED mobile platform.
  Interview data will be analyzed thematically to identify facilitators, barriers, and behavioral impacts related to long-term use.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Beigang Hospital, London, Alabama, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
We will decide if the IPD can be shared before the end of the study.

REFERENCES:
- [Result] Guu TW, Muurling M, Khan Z, Kalafatis C, Aarsland D, Ffytche D, Brem AK. Wearable devices: underrepresentation in the ageing society. Lancet Digit Health. 2023 Jun;5(6):e336-e337. doi: 10.1016/S2589-7500(23)00069-9. No abstract available. PMID 37236695
- [Result] Guu TW, Brem AK, Albertyn CP, Kandangwa P, Aarsland D, Ffytche D. Wrist-worn actigraphy in agitated late-stage dementia patients: A feasibility study on digital inclusion. Alzheimers Dement. 2024 May;20(5):3211-3218. doi: 10.1002/alz.13772. Epub 2024 Mar 18. PMID 38497216